CLINICAL TRIAL: NCT00690443
Title: A Randomized, Double Blind Comparator-controlled, Parallel-group Study to Evaluate the Safety and Efficacy of the Combination of AEGR-733 and Atorvastatin 20 mg vs Atorvastatin Monotherapy in Subjects With Moderate Hypercholesterolemia
Brief Title: Evaluate Safety and Efficacy of AEGR-733 and Atorvastatin vs Atorvastatin Monotherapy in Hypercholesterolemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aegerion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AEGR-733-006
Record Dates: First submitted 2008-05-20; First posted 2008-06-04 (Estimated); Results first posted 2013-02-25 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Hypercholesterolemia
Keywords: Hyperlipidemia
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipidemias | interventions — Atorvastatin; BMS201038

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Active Comparator): 2.5 mg AEGR 733 plus atorvastatin 20 mg weeks 1-4 followed by 5 mg AEGR 733 plus atorvastatin 20 mg weeks 5-8
  Interventions: Drug: AEGR-733
- 1 (Active Comparator): Following 35-day washout + diet run-in, subjects receive atorvastatin 20 mg for 8 wks.
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — atorvastatin 20 mg tablets, daily dosing, for 8 weeks.
  Other Names: Lipitor
  Arms: 1
Drug: AEGR-733 — 2.5 mg AEGR-733 capsules, daily dosing, 4 weeks followed by 5 mg AEGR-733 capsules, daily dosing, 4 weeks
  Arms: 2

SUMMARY:
Evaluate the efficacy of combination therapy AEGR-733 plus atorvastatin 20 mg versus monotherapy on serum lipoproteins over 4 and 8 weeks of therapy. The primary efficacy parameter is percent change in LDL-C after 8 weeks of therapy.

DETAILED DESCRIPTION:
Following a 35-day washout of current lipid-lowering medication (if any) and adherence to a low-fat diet, subjects will receive either atorvastatin 20 mg for 8 weeks, OR AEGR-733 2.5 mg + atorvastatin 20 mg for 4 weeks followed by AEGR-733 5 mg + atorvastatin 20 mg for 4 additional weeks. During the entire study, subjects will be instructed to follow a low-fat/low cholesterol diet and limit alcohol consumption to -/< 1 drink per day.

ELIGIBILITY:
Inclusion Criteria:

* M/F 18-70
* 0-1 risk factor, mean LDL-C -/> 160 and -/< 250 mg/dL (Visit 2 & 3)
* 2+ risk factors, mean LDL-C -/> 130 & -/< 250 mg/dL (Visit 2 & 3)
* Fasting mean TGs -/< 400 mg/dL
* Understanding and compliance of protocol
* sign consent

Exclusion Criteria:

* Females pregnant, lactating, or CBP who have not been using acceptable contraceptive methods over previous 3 months
* Uncontrolled hypertension >180/95 at screening
* Hx of chronic renal insufficiency (serum creatinine > 2.5 mg/dL)
* Hx of liver disease or transaminases > 1.5 X ULN
* Positive for Hepatitis B or C
* Major surgery within past 3 mos
* Cardiac insufficiency defined as functional Class II-Class IV
* Hx of malignancy within previous 5 years
* Participation in another investigational drug study within past 6 wks
* Serious or unstable medical or psychological condition
* Regular alcohol use > 1 drink per day
* Regular consumers of grapefruit juice or medications known to be metabolized by CYP 3A4
* Use of other lipid-lowering meds (washout permitted)
* Acute CVD
* Diabetes Mellitus
* Fasting glucose >110 mg/dL
* BMI -/> 40 kg/m2
* Significant gastrointestinal symptoms such as IBS
* Use of fish oils, niacin, herbal wt. loss products (washout permitted)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2008-05; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Belknap, MD, Study Director — Medical Monitor at Radiant Research
Locations (5):
- United States (5):
  - Linda Murray, DO - Radiant Research, Pinellas Park, Florida
  - Sheila Rodstein, MD, Edina, Minnesota
  - Dennis McCluskey, MD - Radiant Research, Mogadore, Ohio
  - Michele Reynolds, MD, Dallas, Texas
  - William Jennings, MD - Radiant Research, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was performed from 12 May 2008 to 29 Aug 2008. A total of 5 medical clinics participated in the study.
Pre-assignment Details: 5-week run-in period during which patients were to follow a low-fat diet and washout from previous lipid lowering therapies.
Groups:
- Atorvastatin 20 mg: Oral atorvastatin 20 mg for 8 weeks
- Atorvastatin 20 mg + Lomitapide: Oral atorvastatin 20 mg and lomitapide 2.5 mg for 4 weeks, followed by 4 weeks of atorvastatin 20 mg and lomitapide 5 mg
Period: Overall Study
Arm/Group | Atorvastatin 20 mg | Atorvastatin 20 mg + Lomitapide
Started | 23 | 21
Completed | 22 | 19
Not Completed | 1 | 2
Not completed — Adverse Event | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atorvastatin 20 mg | Atorvastatin 20 mg + Lomitapide | Total
Number analyzed (Participants) | 23 | 21 | 44
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.8 (6.22) | 57.8 (8.06) | 58.3 (7.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 24
  Male | 10 | 10 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 18 | 36
  Not Hispanic or Latino | 5 | 3 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 22 | 20 | 42
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: Participants]
  United States | 23 | 21 | 44

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in LDL-C After 8 Weeks of Therapy
Time Frame: Baseline and 8 weeks of treatment
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Atorvastatin 20 mg | Atorvastatin 20 mg + Lomitapide
Number analyzed (Participants) | 22 | 19
Percent Change | -39.6 (14.35) | -49.9 (26.78)

2. Secondary Outcome: Percent Changes in LDL-C at Week 4 + Baseline Serum Lipoproteins (TC, Non-HDL, VLDL, TGs, HDL-C, Apolopoproteins A1 and B), High Sensitivity C-reactive Protein and Change in Body Weight.
Time Frame: Baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Atorvastatin 20 mg | Atorvastatin 20 mg + Lomitapide
Number analyzed (Participants) | 23 | 19
Percent
  Change in LDL-C | -42.5 (12.70) | -51.0 (18.34)
  Change in TC | -31.3 (9.23) | -38.1 (15.38)
  Change in TGs | -21.5 (18.31) | -17.8 (28.32)
  Change in HDL-C | 6.7 (8.07) | -1.9 (10.73)
  Change in non-HDL-C | -39.6 (10.78) | -45.8 (17.68)
  Change in Apo B | -33.6 (10.19) | -37.7 (17.05)
  Change in Apo A-1 | 4.8 (7.53) | -7.8 (8.85)
  Change in hs-CRP | -12.0 (43.21) | 60.5 (187.50)
  Change in body weight | 0.0 (1.38) | -0.7 (1.49)

ADVERSE EVENTS:
Arm/Group | Atorvastatin 20 mg | Atorvastatin 20 mg + Lomitapide
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/21
Other Adverse Events (participants affected / at risk) | 16/23 | 16/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atorvastatin 20 mg (N=23) | Atorvastatin 20 mg + Lomitapide (N=21)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 10 (10)
Flatuence (Gastrointestinal disorders) | 2 (2) | 4 (4)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (3)
Headache (Nervous system disorders) | 2 (2) | 3 (3)
Alanine aminotransferase increased (Investigations) | 0 (0) | 4 (4)
Abdominal distension (Gastrointestinal disorders) | 3 (3) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 3 (3)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (3)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Foot fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Information is unavailable.